CLINICAL TRIAL: NCT03641261
Title: Evaluation of the Feasibility and Effect of Therapeutic Education Sessions Using an Internet Application in Hereditary Ichthyosis
Brief Title: Therapeutic Education Using an Internet Application in Hereditary Ichthyosis
Acronym: e-ETPichtyose
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Toulouse (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: RC31/16/8765
Record Dates: First submitted 2018-06-04; First posted 2018-08-21 (Actual); Last update posted 2024-04-12 (Actual); Status verified 2024-04

CONDITIONS: Ichthyosis
Keywords: Hereditary ichthyosis
MeSH Terms: conditions — Ichthyosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Therapeutic Patient Education program (Experimental): All included patients will follow a Therapeutic Patient Education program dedicated to the hereditary ichthyosis and using a web application, WebIchtyose
  Interventions: Other: Therapeutic patient education program

INTERVENTIONS:
Other: Therapeutic patient education program — WebIchtyose is a specific therapeutic patient education program for patients with hereditary Ichthyosis targeting the problems of each patient by means of a personalized follow-up and a constant interaction between the patient and the educational team
  Other Names: WebIchtyose

SUMMARY:
The main purpose is to evaluate the feasibility (global use) of a therapeutic patient education program using a specific web application in patients with hereditary ichthyosis.

ELIGIBILITY:
Inclusion Criteria:

* Patient with hereditary ichthyosis, according to the classification established during the 2009 consensus conference
* Who has given his informed consent form
* Who is affiliated to a social security system

Exclusion Criteria:

* Patient who has already participated in a therapeutic patient education program for the hereditary ichthyosis
* Unable to connect or use a computer tool
* Impossibility to be present at the only face-to-face session
* Patient who is not available for the collective educational session
* Patient with little or no motivation to follow a therapeutic patient education program (motivation evaluated by the educational team by phone call before inclusion)
* Patient not mastering the French language
* Person under legal protection (guardianship, curators or safeguard of justice)

Ages: 15 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 42 (Actual)
Dates: Start 2018-10-29 (Actual); Primary Completion 2023-02-21 (Actual); Study Completion 2023-02-21 (Actual)

PRIMARY OUTCOMES:
Global use | 6 months
  percentage of patients who have used the "WebIchtyose" application for at least 8 hours during 6 months

SECONDARY OUTCOMES:
Fractional use in each domain (educational sessions) | 6 months
  "WebIchtyose" application use time by the patient for group and individual educational sessions
Fractional use in each domain (continuous educational follow-up) | 6 months
  "WebIchtyose" application use time by the patient for the continuous educational follow-up
Fractional use in each domain (consultation) | 6 months
  "WebIchtyose" application use time by the patient for the consultation of the "Frequently Asked Questions" area and of patient information documents made available on the application
Fractional use in each domain (questionnaires) | 6 months
  "WebIchtyose" application use time by the patient for the filling of the questionnaires
Fractional use in each domain | 6 months
  "WebIchtyose" application use time by the patient for group and individual educational sessions, the continuous educational follow-up, the consultation of the "Frequently Asked Questions" area and of patient information documents made available on the application
Difficulty of individual application registration | Baseline
  Difficulty of registration questionnaire completed for each patient jointly by the patient and the educational team at the end of the face-to-face inclusion visit
Difficulties of use in everyday life by the patient | 6 months
  Questionnaire completed for each patient jointly by the patient at the end of the program
Number of exchanges | 3 months and 5 months
  Number of exchanges necessary between the educational team and the patient to set a date for the conduct of the individual educational sessions
Response time | 6 months
  Response time of the educational team following a request from the patient as part of the educational follow-up
Number of relaunches | 2 months, 4 months and 6 months
  How many times the nurse relaunches the patient to obtain the assessment questionnaires
Number of non-received questionnaires | 2 months, 4 months and 6 months
  Number of non-received questionnaires after relaunch
Number of lost to follow-up patients | 9 months
  Number of lost to follow-up patients
Patient acceptability | 6 months
  Acceptability questionnaire to be completed by the patient
Educational team acceptability | 6 months
  Acceptability questionnaire to be completed by each member of the educational team
Attractiveness | 6 months
  Application attractiveness questionnaire completed by the patient
Quality of life before and after treatment | Inclusion, 6 months and 9 months
  Quality of life questionnaire for hereditary ichthyosis (IQoL-32)
Self-assessment of cutaneous severity | Inclusion and 6 months
  Self-assessment of cutaneous severity according to an analogic visual scale for pain, pruritus, erythema, squama
Knowledge about disease and treatments | Inclusion and 6 months
  Questionnaire of knowledge about disease and treatments
Self-care skills | Inclusion and 6 months
  Questionnaire of self-care skills
Self-esteem | Inclusion and 6 months
  Questionnaire about self-esteem: Rosenberg scale. For each item of the questionnaire, the modality answers are : 1 (totally disagree), 2 (quite disagree), 3 (quite agree) and 4 (totally disagree). The total score (/ 40) is calculated by adding the scores obtained for each item.
Coping scale | Inclusion and 6 months
  Coping with health injuries and problem (Endler 1998). For each item of the questionnaire, the modality answers are: 1 (not at all), 2 (a little), 3 (moderately), 4 (often) and 5 (a lot).The total score (/ 160) is calculated by adding the scores obtained for each item.

CONTACTS AND LOCATIONS:
Overall Officials: Juliette Mazereeuw-Hautier, MD, Principal Investigator — University Hospital, Toulouse
Locations (1):
- CHU Toulouse, Hôpital Larrey, Toulouse, France